CLINICAL TRIAL: NCT04921189
Title: Steroid, Thiamine and Ascorbic Acid During Post-Resuscitation Period for Comatose Out-of-hospital Cardiac Arrest Survivors (STAR) Trial: Multi-center, Randomized, Single-blinded, Controlled Pilot Study
Brief Title: Steroid, Thiamine and Ascorbic Acid for Comatose Out-of-hospital Cardiac Arrest Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Wonju Severance Christian Hospital (Other); Samsung Changwon Hospital (Other); Samsung Medical Center (Other); Chung-Ang University (Other); Hanyang University (Other); Ewha Womans University (Other); Hanil General Hospital (Unknown)
Responsible Party: Principal Investigator, Won Young Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STAR trial
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Postcardiac Arrest Syndrome
Keywords: Postcardiac Arrest Syndrome; Ischemia/reperfusion injury; Neuron-specific enolase; Ascorbic acid; Thiamine; Cortisol
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome; Reperfusion Injury | interventions — Thiamine; Hydrocortisone; Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The combined supplement of Ascorbic acid, Thiamine, and Cortisol (Active Comparator): The combined administration of 3 drugs will be administered through intravenous infusion over 60 min every 12 h for 3 days for the out-of-hospital cardiac arrest survivors treated with targeted temperature management.
  Interventions: Drug: The combined supplement of Ascorbic acid, Thiamine, and Cortisol
- Placebo (Placebo Comparator): An identical volume of 0.9% saline (150mL) administered through intravenous infusion over 60 min every 12 h for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: The combined supplement of Ascorbic acid, Thiamine, and Cortisol — The combined administration of 3 drugs will be mixed in a 50 mL 0.9% saline bag respectively and administered through intravenous infusion over 60 min every 12 h for 3 days.
  1. Ascorbic acid (Ascorbic acid Inj [500mg]®): 50 mg/kg, maximum single dose 3 g, daily dose 6 g
  2. Thiamine (Thiamine hcl inj [50mg]®): 200 mg
  3. Cortisol (Cortisolu inj [100mg]®): 100mg (The main exposure was corticosteroid therapy, defined as the use of systemic corticosteroids. But if unavailable, it could be converted to hydrocortisone-equivalent doses (methylprednisolone 1:5, dexamethasone 1:25, prednisolone 1:4).)
  Other Names: Ascorbic acid; Thiamine hcl; Cortisolu
  Arms: The combined supplement of Ascorbic acid, Thiamine, and Cortisol
Drug: Placebo — An identical volume of 0.9% saline (150mL) administered through intravenous infusion over 60 min every 12 h for 3 days.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The mortality and neurological outcomes among out-of-hospital cardiac arrest survivors have not improved despite the medical advances. The whole body ischemia/reperfusion injuries after cardiac arrest mainly damaged the brain. To improve the neurologic outcome among those patients, additional interventions would be warranted.

The investigators hypothesize that the combined use of cortisol, ascorbic acid (vitamin C), and thiamine during the early post-resuscitation period would attenuate the whole-body ischemia/reperfusion injuries among the out-of-hospital cardiac arrest survivors treated with targeted temperature management.

DETAILED DESCRIPTION:
The mortality and neurological outcomes among the out-of-hospital cardiac arrest survivors are still dismal. In addition, the metabolic and oxidative stress can persist or even worsen at the cellular level after resuscitation, and these whole-body ischemia/reperfusion injuries contribute to multiple organ failure, known as the post-cardiac arrest syndrome. Therefore, additional interventions to reduces the injuries would be warranted.

Cortisol has beneficial antioxidant and anti-apoptotic properties and stabilizes cellular membranes exposed to oxidative stress. It also maintains hemodynamic stability and improves organ function by reducing ischemia/reperfusion injuries.

Thiamine is a cofactor that acts on enzymes essential for glucose metabolism, the generation of adenosine triphosphate, and nicotinamide adenine dinucleotide phosphate production. It assists the cellular metabolisms and attenuates the potential adverse effect of ascorbic acid (vitamin C) by preventing the conversion of ascorbic acid into oxalate. Ascorbic acid is a well-known antioxidant and has anti-inflammatory effects. It acted as an antioxidant defense substance, reducing reactive oxygen species and reactive nitrogen species and improving microcirculation by limiting oxidative injury and endothelial barrier disruption. The theoretical and experimental studies suggested the concomitant use of cortisol, thiamine, and ascorbic acid might have potential treatment synergism for whole-body ischemia/reperfusion injuries after cardiac arrest.

The investigators hypothesize that their combined use during the early post-resuscitation period will reduce the whole-body ischemia/reperfusion injuries, especially the brain, in out-of-hospital cardiac arrest survivors treated with targeted temperature management.

ELIGIBILITY:
Inclusion Criteria:

* An out-of-hospital cardiac arrest survivors treated with targeted temperature management (target between 32 and 36 °C)
* Presumed cardiogenic cause as cardiac arrest

Exclusion Criteria:

* > 12 hours from cardiac arrest to drug or placebo administration
* previous poor neurological status (Cerebral Performance Categories 3 to 5)
* patients who have set limitations on treatment (e.g. patients with a signed do-not-resuscitate order)
* Patients with an underlying terminal-stage disease without an active treatment plan and those who are not expected to survive to discharge
* patients taking at least 1 g/day of vitamin C or receiving intravenous thiamine prior to enrolment
* patients experiencing cardiac arrest prior to enrolment or who are expected to die within 24 h despite best possible treatment, based on the judgement of medical personnel
* pregnant women
* patients with glucose-6-phosphate dehydrogenase deficiency
* patients with a history of hypersensitivity reactions to the trial drugs
* patients with thalassemia
* patients with hyperoxaluria
* patients with cystinuria
* patients with ongoing gout attacks
* patients diagnosed with oxalate renal stones
* patients who do not voluntarily consent to participate in the trial (directly or by legal proxy).

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
the peak neuron-specific enolase level | 48 to 72 hours
  Serum Neuron-Specific Enolase (NSE) level at 48 to 72 hours after resuscitation will measured by enzyme immunoassay, respectively. We will use the peak neuron-specific enolase level.

SECONDARY OUTCOMES:
the delta neuron-specific enolase (NSE) level | at 48, 72 hours
  The delta NSE level is defined as the difference between NSE at 24 hours and the peak NSE between 48 and 72 hours after cardiac arrest.
The delta Sequential Organ Failure Assessment (SOFA) score | at 24, 48, 72 hours
  The delta SOFA is defined as the difference between SOFA admission and SOFA at 72 hours after cardiac arrest. Death within 72 hours will be counted as the maximum SOFA score (24).
30-day Mortality | 30 days
  All-cause death within 30 days
Time to death | 30 days
  The time to death is defined as the duration of survival within 30 days. Survival after 30 days will be counted as 30.
In-hospital mortality | 1 year
  All-cause death during hospitalization
Intensive Care Unit (ICU) stay | The total length of ICU stay will be determined from the date of ICU admission until the patient is discharged from the Intensive Care Unit or the date of death from any cause, assessed up to 1 year after the ﬁrst day of admission.
  1 year
7-day mortality | 7 days
  All-cause death within 7 days
90-day mortality | 90 days
  All-cause death within 90 days
180-day mortality | 180 days
  All-cause death within 180 days
Time to Awakening | 30 days
  Days to neurological recovery, defined as Glasgow Outcome Scale > 13 from cardiac arrest
ICU free day | 14 days
  Days in general ward transferred from ICU within 14 days from admission
Hospital stay | 1 year
  The total hospitalization days
Neurological outcome assessed using Cerebral Performance Category score | at 30, 90, 180 days
  Cerebral Performance Category (CPC) score is defined as follows: CPC 1, Good cerebral performance (normal life); CPC 2, Moderate cerebral disability (disability but independent); CPC 3, Severe cerebral disability (conscious but disabled and dependent); CPC 4, Coma or vegetative state (unconscious); CPC 5, Brain death.
Neurological outcome assessed using the modified Rankin Scale | at 30, 90, 180 days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Won Young Kim, PhD, Study Chair — A
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YJ, Ko BS, Roh YI, Kim YH, Kim WY. Steroid, thiamine, and ascorbic acid during post-resuscitation period for comatose out-of-hospital cardiac arrest survivors (STAR) trial: Protocol for a clinical trial. PLoS One. 2025 Apr 11;20(4):e0319733. doi: 10.1371/journal.pone.0319733. eCollection 2025. PMID 40215244